CLINICAL TRIAL: NCT01331824
Title: Multi-Center Phase 2 Trial of Single-Agent Amrubicin as Second-Line Therapy in Patients With Advanced/Metastatic Refractory Urothelial Carcinoma
Brief Title: Trial of Amrubicin as Second-Line Therapy in Patients With Advanced/Metastatic Refractory Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to a development decision by the funder
Sponsor: Matthew Galsky (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, MD, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 10-1341
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Urothelial Cancer; Chemotherapy; Second-line; Metastatic
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amrubicin (Experimental): 35 mg/m2/day intravenously
  Interventions: Drug: Amrubicin

INTERVENTIONS:
Drug: Amrubicin — Patients will receive 35 mg/m2/day of amrubicin intravenously for 3 consecutive days as the initial dose starting on Day 1 of a 21-day cycle for up to 6 cycles

SUMMARY:
The primary objective of this study is to determine in subjects with metastatic measurable bladder cancer (or urothelial cancers originating elsewhere in the genitourinary tract) who have progressed on 1 prior chemotherapeutic regimen the objective response rate to treatment with amrubicin. The secondary objectives will be to evaluate progression-free survival, survival at 1 year, and the safety of amrubicin as second-line therapy in patients with metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
Multiple small phase II trials exploring a variety of agents as second-line therapy for metastatic urothelial carcinoma have been performed. Overall, the most active of these agents have shown response rates of approximately 10-20% . Currently, there are no FDA approved agents for the second-line treatment of metastatic urothelial carcinoma.

The current study will explore the safety and activity of the novel anthracycline, amrubicin, as second-line chemotherapy in patients with advanced urothelial carcinoma.

The primary objective will be to evaluate the activity (as determined by objective response rate) of amrubicin as second-line chemotherapy in patients with metastatic urothelial carcinoma. The secondary objectives will be to evaluate progression-free survival, survival at 1 year, and the safety of amrubicin as second-line therapy in patients with metastatic urothelial carcinoma.

Subjects will receive amrubicin IV daily x 3 days, every 21-days, with prophylactic granulocyte colony stimulating factor. This 21-day time period is referred to as a cycle. Subjects will undergo repeat computed tomography (CT) scans after every 2 cycles. In the absence of progressive cancer, or prohibitive side effects, subjects will receive up to 6 cycles of treatment with amrubicin.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age > 18 years
3. Karnofsky performance status of ≥ 80%
4. Histological or cytological proof of transitional cell carcinoma of the urothelial tract. The primary site may include: urethra, bladder, ureters, and renal pelvis.
5. Progressive advanced/metastatic disease despite prior chemotherapy:

   * Patients may have received one prior chemotherapy regimen.
   * Prior chemotherapy may have been administered in the perioperative setting (neoadjuvant or adjuvant) or 1st line metastatic setting.
6. Measurable disease according to RECIST 1.1
7. Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 8 weeks after treatment discontinuation.
8. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.
9. Adequate organ function including the following:

   * Adequate bone marrow reserve: absolute neutrophil count (segmented and bands) (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, and hemoglobin ≥ 9 mg/L,
   * Hepatic: bilirubin ≤ 1.5 x the upper limit of normal (ULN), ALT and AST ≤ 3.0 x ULN (or ≤ 5.0 x ULN in the presence of hepatic metastases)
   * Renal: serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 60 mL/min,
   * Cardiac: Left ventricular ejection fraction (LVEF) ≥ 50% or ≥ the lower limit of the institutional normal by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA);

Exclusion Criteria:

1. Has had major surgery within 30 days of starting study treatment.
2. Has active CNS metastases. Subjects with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis.
3. Has a history of a prior malignancy with the exception of the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, clinically localized prostate cancer treated with definitive local therapy and without evidence of recurrent disease and without the need for androgen deprivation therapy, or other cancer for which the subject has been disease-free for at least 5 years.
4. Has had treatment with another anticancer agent or investigational agent within 30 days prior to being registered for protocol therapy.
5. Has had prior radiation therapy to > 25% of the bone marrow.

   * NOTE: No radiation therapy within 30 days prior to being registered for protocol therapy.
6. Has a clinically significant infection as judged by the treating investigator.
7. Pregnant or nursing females.
8. Patients with known history of seropositive human immunodeficiency virus (HIV) or patients who are receiving immunosuppressive medications that would, in the opinion of the investigator, increase the risk of serious neutropenic complications.
9. History of congestive heart failure
10. History of recent myocardial infarction
11. History of interstitial lung disease, pulmonary fibrosis or symptomatic pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-02; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Amrubicin: Patients with progressive metastatic urothelial cancer despite first-line chemotherapy. Amrubicin was initially administered at a dose of 40 mg/m2/day daily x 3 every 21-days and the dose was subsequently reduced to 35 mg/m2/day daily x 3 every 21-days.
Period: Overall Study
Arm/Group | Amrubicin
Started | 22
Completed | 9
Not Completed | 13
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Disease Progression | 9
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Amrubicin
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 65 [58 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 18
Primary Site [Number; unit: participants]
  Bladder | 16
  Renal Pelvis | 3
  Urethra | 3
Prior "first-line" treatment [Number; unit: participants]
  Neoadjuvant | 4
  Adjuvant | 4
  Metastatic | 14
First-line chemotherapy regimen [Number; unit: participants]
  Gemcitabine + carboplatin | 7
  Gemcitabine + cisplatin | 12
  Gemcitabine + cisplatin + dovitinib | 1
  Gemcitabine + cisplatin + ipilimumab | 1
  Gemcitabine + doxorubicin + paclitaxel | 1
Bellmunt prognostic factors [Number; unit: participants] — The significant prognostic factors were as follows: hemoglobin level more than 10 g/dL, ECOG PS less than 1, absence of liver metastases, metastasis restricted to one organ, and AST and AP levels in the normal range.
  participants
    0 poor prognostic factors | 3
    1 poor prognostic factors | 10
    2 poor prognostic factors | 6
    3 poor prognostic factors | 3
Median time from prior chemotherapy [Median (Full Range); unit: months] | 6.8 [1.4 to 34.2]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Description: Response to treatment based on tumor measurements via CT chest, abdomen, and pelvis for restaging after every 2 cycles.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 6 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Amrubicin
Number analyzed (Participants) | 22
percentage of participants
  Partial response | 13.6 [0 to 28]
  Stable disease | 54.5 [33.7 to 75.3]

2. Secondary Outcome: Progression-free Survival
Description: The median progression-free survival
  After the last dose of Amrubicin, patients will have follow-up every 3 months with a repeat CT scan of the chest, abdomen, and pelvis until the time of disease progression is documented.
Time Frame: Every 3 months post Amrubicin administration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amrubicin
Number analyzed (Participants) | 22
months | 3.4 [2.1 to 4.8]

3. Secondary Outcome: Overall Survival
Description: The median overall survival
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Amrubicin
Number analyzed (Participants) | 22
months | 7.2 [4.2 to 10.1]

4. Secondary Outcome: Safety as Measured by the Frequency and Type of Adverse Events as Per the Common Terminology for Adverse Events (CTCAE) Version 4.0.
Description: Types of adverse events listed in Adverse Event Section
Time Frame: Day 1 of each treatment cycle; and 21 days after the last dose of amrubicin
Measure: Number; unit: adverse events
Arm/Group | Amrubicin
Number analyzed (Participants) | 22
adverse events | 117

ADVERSE EVENTS:
Arm/Group | Amrubicin
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amrubicin (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amrubicin (N=22)
Alopecia (Skin and subcutaneous tissue disorders) | 13
Anemia (Blood and lymphatic system disorders) | 10
Anorexia (General disorders) | 6
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Conjunctival irritation (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Creatinine increase (Renal and urinary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 13
Fever (General disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Mucositis (Injury, poisoning and procedural complications) | 9
Nausea (General disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 4
Taste alteration (General disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Urinary frequency (Renal and urinary disorders) | 1
Vomiting (General disorders) | 7
Weakness (Nervous system disorders) | 2
Weight loss (General disorders) | 3

LIMITATIONS AND CAVEATS:
The trial was terminated prematurely due to the results of a phase 3 study seeking registration for amrubicin in small cell lung cancer in the United States, leading the industry funder to discontinue further clinical development of amrubicin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes